CLINICAL TRIAL: NCT01797861
Title: A Prospective Randomized Controlled Multicentre Trial Comparing Half-dose Photodynamic Therapy (PDT) With High-density Subthreshold Micropulse Laser Treatment in Patients With Chronic Central Serous Chorioretinopathy (CSC)
Brief Title: Prospective Randomized Controlled Treatment Trial for Chronic Central Serous Chorioretinopathy
Acronym: PLACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Cologne (Other); University of Oxford (Other); Leiden University Medical Center (Other); University Hospital, Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLACE
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2016-04

CONDITIONS: Chronic Central Serous Chorioretinopathy
Keywords: chronic central serous chorioretinopathy; photodynamic therapy; micropulse laser
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Half-dose photodynamic therapy (PDT) (Active Comparator): In the PDT treatment arm, all patients will receive an intravenous drip through which half-dose (3 mg/m2) verteporfin (Visudyne ®) is administered, with an infusion time of 10 minutes. At 15 minutes after the start of the infusion, PDT laser treatment is performed with standard 50 J/cm2 fluency, a wavelength of 689 nm, and a treatment duration of 83 seconds.
  If there still is subretinal fluid on OCT scan at Evaluation Visit 1 (6-8 weeks after Treatment Visit 1 / the first treatment with half-dose PDT), a second treatment with half-dose PDT will be performed (Treatment Visit 2).
  Interventions: Procedure: Half-dose photodynamic therapy (PDT)
- Micropulse laser (ML) treatment (Active Comparator): ML treatment with an 810 nm diode laser will be performed of the areas identified on mid-phase ICG angiography. Multiple laser spots will be applied, covering the leakage area on mid-phase ICG angiography. The area(s) that has to be treated is determined based on those hyperfluorescent area(s) on mid-phase (approximately 10 minutes) ICG-angiography that correspond to subretinal fluid accumulation in the macula on the OCT scan and hyperfluorescent "hot spots" on the mid-phase (3 minutes) fluorescein angiogram.
  If there still is subretinal fluid on OCT scan at Evaluation Visit 1 (6-8 weeks after Treatment Visit 1 / the first ML treatment), a second ML treatment will be performed (Treatment Visit 2).
  Interventions: Procedure: Micropulse laser (ML) treatment

INTERVENTIONS:
Procedure: Half-dose photodynamic therapy (PDT) — At exactly 15 minutes after the start of the half-dose verteporfin infusion, the PDT treatment will take place. The area that has to be treated with the PDT laser is determined based on those hyperfluorescent area(s) on mid-phase (approximately 10 minutes) ICG-angiography that correspond to subretinal fluid accumulation in the macula on the OCT scan and hyperfluorescent "hot spots" on the mid-phase (approximately 3 minutes) fluorescein angiogram. The spot size will be defined based on diameter of the hyperfluorescent area on ICG angiography plus 1mm. The treatment is performed with standard fluency (50 J/cm2), a PDT laser wavelength of 689 nm, and a standard treatment duration of 83 seconds.
  Arms: Half-dose photodynamic therapy (PDT)
Procedure: Micropulse laser (ML) treatment — The following ML treatment settings will be used: a power of 1800 mW*, a duty cycle of 5%, frequency of 500 Hz, exposure time of 0.2 s per spot, spot size: 125 µm, minimal distance of spot from fovea: 500 µm.
  * Subthreshold treatment is desired, meaning that no visible reaction due to laser treatment has to be seen in the retina. In virtually all patients, a power of 1800 mW wil not produce a visible discoloration of the retina after application of a laser spot with the aforementioned settings. If retinal discoloration is seen at a power of 1800 mW the power will be reduced with steps of 300 mW until there is no visible reaction. The first laser "test" spot will always be applied just outside the macular area.
  Arms: Micropulse laser (ML) treatment

SUMMARY:
Chronic central serous chorioretinopathy (CSC) is a relatively frequent eye disease that often occurs in patients in the professionally active age range. In this disease, there is pooling of fluid under the central retina (the macula). This specific form of macular degeneration can cause permanent vision loss, image distortion, loss of color and contrast vision due to this fluid under the retina. An early diagnosis and treatment may improve the visual outcome and quality of life. To date there is no international consensus on the optimal treatment of chronic CSC. Many retrospective studies suggest that treatment with photodynamic therapy (PDT) is effective in chronic CSC. Micropulse laser (ML) therapy may also be effective in this disease.

The proposed study is the first prospective randomized controlled trial in chronic CSC. In this study, participants with chronic CSC will be randomized into two treatment groups, PDT or ML treatment. The trial is a superiority study, because retrospective studies suggest that PDT treatment may be more effective than ML treatment. Therefore, PDT treatment is challenged against ML treatment.

The null hypothesis of the study is that PDT treatment is more effective than ML treatment in patients with active chronic CSC. The alternative hypothesis is that PDT treatment is not more effective than ML treatment in these patients.

Treatment success will not only be based on anatomical improvement, but also on functional endpoints, which are most important from a patient's perspective.

The study will take place in five large tertiary referral university hospitals in Europe that have extensive experience with conducting clinical trials (in Nijmegen, the Netherlands; Cologne, Germany; Leiden, the Netherlands; Oxford, United Kingdom; and Paris, France). Each of these centers has confirmed sufficient funding to conduct the research. The study will last max. 8 months per participant. Each participant will come for 5 (in the case of 1 treatment) or 7 visits (in the case of 2 treatments). Study evaluations will be mostly part of regular clinical care. The whole study will last for max. 24 months.

DETAILED DESCRIPTION:
PURPOSE AND DESIGN There is no international consensus on the optimal treatment protocol of chronic CSC. Nevertheless, photodynamic therapy (PDT) has emerged as the treatment of choice in many centres worldwide. PDT uses a photosensitive drug, verteporfin (Visudyne®), that is administered once intravenously before treatment with a specific type of laser. PDT treatment has been developed originally as treatment for another form of macular degeneration, age-related macular degeneration, on which there are extensive data available. There are several other retinal diseases for which PDT with verteporfin is successfully used as an off-label treatment. The use of PDT treatment in chronic CSC is based on the high rate of anatomic success, the increase of visual acuity, the improvement in retinal sensitivity, and an excellent safety profile reported in many retrospective studies. The PDT strategies that are generally used are either with half the dose of verteporfin (Visudyne®) and full fluence (energy) of laser treatment, half the fluence level and the full dose of verteporfin, or half the treatment time using the full dose of verteporfin and full fluence, as compared to the original protocol that was used for neovascular age-related macular degeneration. These PDT strategies that use either half-dose of half-fluence treatment have been developed because a combination of the dosage and fluence that was originally used for the treatment of neovascular age-related macular degeneration showed a higher risk of developing choroidal ischemia and retinal atrophic changes. The half-dose and half-fluence PDT strategies, however, have been shown to be safe and effective in relatively large retrospective studies and one non-controlled non-randomized prospective study by Chan et al. in chronic CSC patients with sufficient follow-up periods.

Therefore, tailoring the therapy to obtain the maximal treatment effect with minimal toxicity is essential in treating patients with CSC. By reducing the dose of verteporfin, studies have demonstrated that the potential retinal damage caused by PDT can be minimized while the photodynamic effects in inducing choroidal vasculature changes required for treating CSC remain sufficient. We have chosen for half-dose because this "safety-enhanced" protocol appeared to be one of the safest and effective treatment options in patients with active chronic CSC.

PDT will be compared with micropulse laser (ML) treatment as a control arm, and not with sham or conventional laser treatment, for a number of reasons. First, sham (no treatment) was studied by Chan et al. who showed a large difference in anatomic outcome (complete resolution of subretinal fluid) and functional outcome (visual acuity) between the half-dose PDT and placebo group in the acute form of CSC, which often resolves spontaneously after a few weeks in contrast to chronic CSC. As it is well-established that prolonged leakage of subretinal fluid under the macula due to chronic CSC may lead to permanent visual loss, it is not desirable to compare half-dose PDT treatment with sham. Apart from these ethical considerations to refrain from comparing with sham, adding a third sham study arm would require an extra amount of study patients that would complicate the recruitment process. The treatment of CSC with ML treatment has been shown to be effective and safe in retrospective studies in 41-58% of patients. The safety and efficacy of ML treatment has also been shown in various other retinal diseases. In contrast, it has been shown that conventional laser treatment of focal leakage point on fluorescein angiography in CSC does not result in a better visual outcome. Also, conventional laser treatment has a higher risk of complications then ML and PDT, including visual loss, scotoma, decreased color vision, decreased contrast sensitivity, and choroidal neovascularization.

The proposed study is a superiority study, as retrospective studies suggest that the rate of anatomical and functional success of half-dose PDT treatment might be higher than ML treatment. However, none of these previous studies on half-dose PDT and ML treatment were prospective, randomized, as well as controlled. Therefore, we have chosen to challenge the half-dose PDT treatment arm against a treatment arm of ML treatment.

The number of visits and examinations have been reduced to a minimum, and conform to standard clinical care as much as possible. Extra examinations include a more extensive visual acuity measurement, microperimetry, and a questionnaire. These extra examinations are required to evaluate the functional vision-related endpoints of the study. Care will be taken to plan all examinations on the same day as much as possible.

RECRUITMENT AND CONSENT Patients will be informed about the treatment options for their eye disease that are currently available. Study investigators will obtain consent for participation in the study, but consent for currently available treatments outside the study will be obtained by medical and nursing staff as would be done routinely. Written and verbal versions of the participant information and informed consent will be presented to the participants, detailing the exact nature of the study, the implications and constraints of the protocol, the known side effects, and any risks involved in taking part. It will be clearly stated that the participant is free to withdraw from the study at any time for any reason without prejudice to future care, and with no obligation to give the reason for withdrawal. Care will be taken to avoid coercion and undue influence of the "recruiter" on the potential participant.

The potential participant will be allowed as much time as wished to consider the information, and the opportunity to question the Investigator, their General Practitioner or other independent parties to decide whether they will participate in the study.

CONFIDENTIALITY The source documents and participants' Case Report Form (CRF) data will always remain in the study centre in which the patient is treated (either Oxford, Cologne, Paris, or Nijmegen). No person-identifiable information will be used unless it is absolutely necessary. The trial staff will ensure that the participants' anonymity is maintained. The participants will be identified only by initials and a participants identification number on the CRF and the electronic database. All documents will be stored securely and only accessible by trial staff and authorised personnel. The study will comply with the Data Protection Act which requires data to be anonymized as soon as it is practical to do so. Anonymized data will be entered into a purpose-built digital database that is maintained by a contract research organisation, the Clinical Research Centre Nijmegen (www.crcn.nl), which is affiliated with the coordinating academic centre, the Institute of Ophthalmology of the Radboud University Nijmegen Medical Centre in Nijmegen the Netherlands.

ELIGIBILITY:
INCLUSION CRITERIA:

* male and female patients ≥ 18 years of age who are able to give written informed consent
* active chronic central serous chorioretinopathy
* subjective visual loss > 6 weeks, interpreted as onset of active disease
* subretinal fluid that includes the fovea on OCT scanning at Baseline Examination.

Please NOTE: Subretinal fluid does not have to include fovea on OCT to be eligible for treatment at Control Visit 1, as long as there is persistent subretinal fluid in the macula, which is interpreted as persistently active disease (see 5.7 "Retreatment criteria and considerations").

* hyperfluorescent areas on ICG angiography
* ≥1 ill-defined hyperfluorescent leakage areas on fluorescein angiography with retinal pigment epithelial window defect(s) that are compatible with chronic CSC

EXCLUSION CRITERIA:

The participant may not enter the study if ANY of the following apply:

* any previous treatments for active CSC in the study eye
* current treatment with corticosteroids (topical or systemic), or anticipated start of corticosteroid treatment within the first 7-8 months from the start of the trial period
* evidence of other diagnosis that can explain serous subretinal fluid or visual loss
* BCVA < 20/200 (Snellen equivalent)
* profound chorioretinal atrophy in central macular area on ophthalmoscopy and OCT
* myopia > 6 dioptres
* visual loss and/or serous detachment on OCT < 6 weeks
* continuous and/or progressive visual loss > 18 months or serous detachment on OCT > 18 months
* no hyperfluorescence on ICG angiography
* intraretinal edema on OCT
* (relative) contraindications for PDT treatment (pregnancy, porphyria, severely disturbed liver function). Pregnancy will not be routinely tested in female patients, but the possibility of pregnancy will be discussed during eligibility screening
* (relative) contraindications for fluorescein angiography or ICG angiography (known allergies especially against shellfish, previous reactions)
* Soft drusen in treated eye or fellow eye, signs of choroidal neovascularization on ophthalmoscopy and/or fluorescein angiography/indocyanine green angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Absence of subretinal fluid on OCT scan | 6-8 weeks after treatment
  The primary endpoint of this study is to assess if there is a difference between the efficacy of half-dose photodynamic therapy treatment versus micropulse laser treatment in patients with chronic central serous chorioretinopathy. The assessment of this efficacy will be based on the anatomical effect on optical coherence tomography (OCT): absence of subretinal fluid versus persistent subretinal fluid, 6-8 weeks after treatment. After all, the absence or presence of fluid under the retina on the OCT scan is a direct reflection of the activity of the disease in these patients.

SECONDARY OUTCOMES:
Best-corrected visual acuity | 6-8 weeks and 7-8 months after Treatment Visit 1
  As secondary endpoints, we will mainly look at three parameters that reflect the patient's vision-related functioning. These three parameters are: a standardized measurement of best-corrected visual acuity (BCVA) according to the Early Treatment of Diabetic Retinopathy Study (ETDRS) standards, a standardized measurement of sensitivity of the macula with microperimetry, and standardized assessment of the patient's vision-related quality of life using a validated questionnaire, the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25).
  The secondary endpoint with regard to BCVA that will be assessed as a reflection of functional improvement after treatment includes:
  * Mean change from baseline in ETDRS BCVA in the study eye at 6-8 weeks after Treatment Visit 1 and at 7-8 months after Treatment Visit 1
  * Mean change from Evaluation Visit 1 in ETDRS BCVA in the study eye at final evaluation (7-8 months after Treatment Visit 1)

OTHER OUTCOMES:
Macular sensitivity on microperimetry | 6-8 weeks and 7-8 months after Treatment Visit 1
  As secondary endpoints, we will mainly look at three parameters that reflect the patient's vision-related functioning. These three parameters are: a standardized measurement of best-corrected visual acuity (BCVA) according to the Early Treatment of Diabetic Retinopathy Study (ETDRS) standards, a standardized measurement of sensitivity of the macula with microperimetry, and standardized assessment of the patient's vision-related quality of life using a validated questionnaire, the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25).
  The secondary endpoint with regard to macular sensitivity that will be assessed as a reflection of functional improvement after treatment includes:
  - Mean change from baseline in retinal sensitivity on microperimetry in the study eye at 6-8 weeks after Treatment Visit 1 and at 7-8 months after Treatment Visit 1 among the two treatment modalities
Vision-related quality of life as reported on the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) | 6-8 weeks and 7-8 months after Treatment Visit 1
  As secondary endpoints, we will mainly look at three parameters that reflect the patient's vision-related functioning. These three parameters are: a standardized measurement of best-corrected visual acuity (BCVA) according to the Early Treatment of Diabetic Retinopathy Study (ETDRS) standards, a standardized measurement of sensitivity of the macula with microperimetry, and standardized assessment of the patient's vision-related quality of life using a validated questionnaire, the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25).
  The secondary endpoint with regard to vision-related quality of life that will be assessed as a reflection of functional improvement after treatment includes:
  - Mean change from baseline in the NEI VFQ-25 questionnaire at 6-8 weeks after Treatment Visit 1 and at 7-8 months after Treatment Visit 1 among the two treatment modalities
Number of second treatments | 7-8 months after Treatment Visit 1
  Another secondary endpoint concerns the number patients in each treatment arm who required a second treatment in an attempt to achieve an absence of subretinal fluid under the retina on OCT at 7-8 months after Treatment Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Camiel JF Boon, MD PhD FEBO, Study Chair — Leiden University Medical Center & Radboud University Nijmegen Medical Center; Carel B Hoyng, MD PhD, Principal Investigator — Radboud University Medical Center; Sacha Fauser, MD PhD, Principal Investigator — Cologne University Eye Clinic; Giuseppe Querques, MD PhD, Principal Investigator — Creteil University Eye Clinic, Paris; Susan M Downes, MD FRCOphth, Principal Investigator — Oxford Eye Hospital; Robert E MacLaren, PhD FRCO, Principal Investigator — University of Oxford
Locations (5):
- Creteil University Eye Clinic, Paris, France
- Cologne University Eye Clinic, Cologne, Germany
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Radboud University Nijmegen Medical Centre, Institute of Ophthalmology, Nijmegen
- Oxford University Eye Hospital, John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feenstra HMA, Hahn LC, van Rijssen TJ, Tsonaka R, Breukink MB, Keunen JEE, Peters PJH, Dijkman G, Souied EH, MacLaren RE, Querques G, Downes SM, Fauser S, Hoyng CB, van Dijk EHC, Boon CJF. EFFICACY OF HALF-DOSE PHOTODYNAMIC THERAPY VERSUS HIGH-DENSITY SUBTHRESHOLD MICROPULSE LASER FOR TREATING PIGMENT EPITHELIAL DETACHMENTS IN CHRONIC CENTRAL SEROUS CHORIORETINOPATHY. Retina. 2022 Apr 1;42(4):721-729. doi: 10.1097/IAE.0000000000003363. PMID 34864802
- [Derived] Pfau M, van Dijk EHC, van Rijssen TJ, Schmitz-Valckenberg S, Holz FG, Fleckenstein M, Boon CJF. Estimation of current and post-treatment retinal function in chronic central serous chorioretinopathy using artificial intelligence. Sci Rep. 2021 Oct 14;11(1):20446. doi: 10.1038/s41598-021-99977-4. PMID 34650220
- [Derived] van Rijssen TJ, Hahn LC, van Dijk EHC, Tsonaka R, Scholz P, Breukink MB, Blanco-Garavito R, Souied EH, Keunen JEE, MacLaren RE, Querques G, Fauser S, Downes SM, Hoyng CB, Boon CJF. RESPONSE OF CHOROIDAL ABNORMALITIES TO PHOTODYNAMIC THERAPY VERSUS MICROPULSE LASER IN CHRONIC CENTRAL SEROUS CHORIORETINOPATHY: Place Trial Report No. 4. Retina. 2021 Oct 1;41(10):2122-2131. doi: 10.1097/IAE.0000000000003157. PMID 34543244
- [Derived] van Dijk EHC, Fauser S, Breukink MB, Blanco-Garavito R, Groenewoud JMM, Keunen JEE, Peters PJH, Dijkman G, Souied EH, MacLaren RE, Querques G, Downes SM, Hoyng CB, Boon CJF. Half-Dose Photodynamic Therapy versus High-Density Subthreshold Micropulse Laser Treatment in Patients with Chronic Central Serous Chorioretinopathy: The PLACE Trial. Ophthalmology. 2018 Oct;125(10):1547-1555. doi: 10.1016/j.ophtha.2018.04.021. Epub 2018 Jun 14. PMID 29776672
- [Derived] Breukink MB, Mohr JK, Ossewaarde-van Norel A, den Hollander AI, Keunen JE, Hoyng CB, Boon CJ. Half-dose photodynamic therapy followed by diode micropulse laser therapy as treatment for chronic central serous chorioretinopathy: evaluation of a prospective treatment protocol. Acta Ophthalmol. 2016 Mar;94(2):187-97. doi: 10.1111/aos.12938. Epub 2015 Dec 15. PMID 26670630
- [Derived] Breukink MB, Downes SM, Querques G, van Dijk EHC, den Hollander AI, Blanco-Garavito R, Keunen JEE, Souied EH, MacLaren RE, Hoyng CB, Fauser S, Boon CJF. Comparing half-dose photodynamic therapy with high-density subthreshold micropulse laser treatment in patients with chronic central serous chorioretinopathy (the PLACE trial): study protocol for a randomized controlled trial. Trials. 2015 Sep 21;16:419. doi: 10.1186/s13063-015-0939-z. PMID 26390920